CLINICAL TRIAL: NCT03695055
Title: Maintenance Therapy After Autologous Hematopoietic Stem Cell Transplantation in High-risk Aggressive Lymphoma
Brief Title: Maintenance Therapy Post-HSCT in High-risk Aggressive Lymphoma
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Ting YANG, Prof.M.D.Ph.D, Fujian Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Lym-SCT-001
Record Dates: First submitted 2018-10-02; First posted 2018-10-03 (Actual); Last update posted 2018-10-03 (Actual); Status verified 2018-10

CONDITIONS: High-risk Aggressive Lymphoma After Auto-HSCT

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1 (Experimental): Rituximab maintenance
  Interventions: Drug: Maintenance therapy post-HSCT
- Arm 2 (Active Comparator): DPP/DCEP-G alternation regimen
  Interventions: Drug: Maintenance therapy post-HSCT
- Arm 3 (No Intervention)

INTERVENTIONS:
Drug: Maintenance therapy post-HSCT — Rituximab vs DPP/DCEP-G vs observation
  Arms: Arm 1; Arm 2

SUMMARY:
Relapse after autologous hematopoietic stem cell transplantation (ASCT) is still challenging for high-risk aggressive lymphoma. This study was to investigate the efficacy and safety of maintenance therapy post-ASCT.

ELIGIBILITY:
Inclusion Criteria:

* Age 14-70 years
* High-risk aggressive lymphoma underwent auto-HSCT
* Presence of 2 or more signs of unfavorable prognosis (IPI 2-4)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
* Adequate hematological function
* Offer informed consent

Exclusion Criteria:

* Concomitant other cancer
* Congestive heart failure, unstable angina, severe cardiac arrhythmias and conduction disturbances, myocardial infarction
* Renal insufficiency (serum creatinine greater than 0.2 mmol/L) (except cases with specific kidney infiltration, urinary tract compression by tumor conglomerate or presence of uric acid nephropathy due to massive cytolysis syndrome)
* Liver failure (except cases with liver tumor infiltration), acute hepatitis or active phase of chronic hepatitis B or C with serum bilirubin greater than 1.5 standards, alanine aminotransferase (ALT) and aspartate aminotransferase (AST) greater than 3 standards, prothrombin index less than 70%
* Severe pneumonia (except cases with specific lungs infiltration), accompanied by respiratory failure (dyspnea > 30 in min., hypoxemia less than 70 mm Hg, when it is impossible to compensate situation in 2-3 days)
* Severe mental disorders (delusions, severe depressive syndrome and other manifestations of productive symptoms) not related with specific infiltration of central nervous system
* Pregnancy

Ages: 14 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-01 (Actual); Primary Completion 2020-01 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Relapse rate | 2 years

SECONDARY OUTCOMES:
Overall survival | 2 years
Treatment-related mortality | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian Medical University Union Hospital, Fuzhou, Fujian, China